CLINICAL TRIAL: NCT06217107
Title: [2069264-1] Wellness & Workforce Solution for Lupus and Lupus Nephritis / Janssen Clinical Investigator Initiated Study
Brief Title: Wellness & Workforce Solution for Lupus/Lupus Nephritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Morehouse School of Medicine (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NOPRODSLE4002
Record Dates: First submitted 2023-12-08; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Lupus Nephritis
Keywords: Lupus; Lupus Nephritis; Health360x; Behavioral Intervention; Health coach; Health Literacy
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C3 Coach plus H360x (Experimental): Arm 1 will have 80 participants who will receive four weekly goal setting sessions with coach consisting of 45 min-1 hour recorded sessions. They will then receive another 4 sessions every 2 weeks, followed by three monthly goal setting sessions. Baseline surveys will be collected, in addition to surveys taken at 3 and 6 months.
  Interventions: Behavioral: Health360x app; Behavioral: Culturally congruent coaching
- C3 Coach plus Health360x and micro-learning (Active Comparator): Arm 2 will have 80 participants who will receive four weekly goal setting sessions with coach consisting of 45 min-1 hour recorded sessions, in addition to periodic micro-learning content delivered via an online technology platform. They will then receive another 4 sessions every 2 weeks, followed by three monthly goal setting sessions. Baseline surveys will be collected, in addition to surveys taken at 3 and 6 months. This arm will have learning augmented by micro-learning to test effectiveness in enhancing engagement and promoting retention of educational content.
  Interventions: Behavioral: Micro-learning content; Behavioral: Health360x app; Behavioral: Culturally congruent coaching

INTERVENTIONS:
Behavioral: Micro-learning content — This is a series of modules designed to provide disease education, additional communication through 'push notifications,' promote self-management, and medication adherence in women of color with lupus and lupus nephritis. Leveraging technology, this program is asynchronous, promotes engagement and retention of information through micro-learning, and allows the investigators to better understand patient experiences beyond structured surveys by capturing what is happening in the patient-coach relationship.
  Arms: C3 Coach plus Health360x and micro-learning
Behavioral: Health360x app — The coach and participant will use problem-solving tools embedded in Health360x to map out potential barriers to goal attainment and create goal action plans. This application has the potential to help improve health-related quality of life, and reduce morbidity and mortality associated with Lupus. The intervention also tests the role of health coaches in the lupus ecosystem. The potential economic gain and impact on more extant social determinants of health can create long ranging benefits on the health and wellbeing of the community.
Behavioral: Culturally congruent coaching — The coaching process includes specified visits over the course of our proposed 6-month intervention. These visits will occur remotely using HIPAA compliant video conferencing tools or in person when it is safe and convenient to meet in person. Overall, the coaches will work with Lupus patients to facilitate experiential learning, improve functioning and performance in the context of working towards specific goals.

SUMMARY:
The investigators will test the hypothesis that culturally congruent coaching delivered via a technology application (Health360x) will improve the persistent disparities observed among women of color with lupus or lupus nephritis by addressing underlying psychosocial barriers to behavioral change.

DETAILED DESCRIPTION:
The investigators' proposed intervention combines technology with culturally congruent coaching (C3) to increase access and engagement of women of color with lupus through remote instruction. The investigators will test the hypothesis that culturally congruent coaching delivered via a technology application (Health360x) will improve the persistent disparities observed among women of color with lupus or lupus nephritis by addressing underlying psychosocial barriers to behavioral change. The investigators will attain this by connecting patients to extensively trained coaches who have lived experiences that clinicians and providers often lack. These shared social and cultural experiences breeds trust and allows for more open communication that the coach can use to provide more appropriate guidance. Leveraging technology, the investigators' program is asynchronous, promotes engagement and retention of information through micro-learning, and allows the investigators to better understand patient experiences beyond structured surveys by capturing what is happening in the patient-coach relationship.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. females ; Age over 18yo
4. Self-reported diagnosis of Lupus or Lupus Nephritis, or documented diagnosis of Lupus or Lupus Nephritis
5. Willingness to adhere to the study intervention regimen
6. Access to necessary resources for participating in a technology-based intervention (i.e., computer, smart-phone, internet access)
7. Not currently practicing self-management behaviors and have not participated in a class or program on self-management behavior within the last 12 months

Adult women with lupus and lupus nephritis will be enrolled in the study. Eligibility: Adult women with lupus and lupus nephritis who are able to consent and participate in self-management support training. Access to the internet is required for this intervention. Ability to read English is required because all the materials are currently in English.

Coaches must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for duration of study
3. Women of color with lupus or lupus nephritis with desire to help others
4. Ability to communicate in English
5. Secure access to Internet
6. Private space for conducting participant visits
7. Ability to use internet-based platform

Exclusion Criteria:

-Potential participants and coaches who are unable to speak or read English, access the internet, or complete data collection activities will be ineligible for participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women of color with lupus and lupus nephritis
Enrollment: 160 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
engagement | Baseline, 3, 6 months
  frequency counts of app usage and patterns of usage will be combined to report application usage data
goal attainment | Baseline, 6 months
  Health360x application usage data

SECONDARY OUTCOMES:
change in systolic and diastolic blood pressure (mmHg) | Baseline, 3, 6 months
  Wireless or Universal Serial Bus enabled patient data upload
change in diet | Baseline, 6 months
  manual entry
change in blood glucose (mg/dL) | Baseline, 3, 6 months
  Wireless or Universal Serial Bus enabled patient uploads
change in total distance walked daily | Baseline, 3, 6 months
  Wireless or Universal Serial Bus enabled patient uploads
Health related quality of life | Baseline, 3, 6 months
  Health related quality of life measure in adult lupus 34 items across 8 domains (physical health, emotional health, body image, pain, planning, fatigue, intimate relationships, and burden to others); A mean raw score is transformed to scores ranging from 0 (worst health related quality of life) to 100 (best health related quality of life)
Fatigue | Baseline, 3, 6 months
  Functional assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-Fatigue); 13-item patient-reported outcome instrument (PRO) that was designed to assess fatigue-related symptoms and impacts on daily functioning; Item scores can range from 0 ("not at all") to 4 ("very much"), and the total score from 0 to 52; lower scores indicate greater fatigue
Stress Management | Baseline, 3, 6 months
  Perceived Stress Scale-4; Individual scores on the Perceived Stress Scale can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Pain will be measured by Brief Pain Inventory - Short Form (BPI-SF) | Baseline, 3, 6 months
  Brief Pain Inventory - Short Form (BPI-SF); Patients are asked to rate their current symptoms, their average experiences of pain, and the minimum and maximum intensities of their symptoms on scales that range from 0 to 10. A total pain severity score can be found by averaging these items or a single item can be treated as the primary outcome measure. A score relating to impact on daily life can be calculated by averaging scores on each of the seven items, which also use scales from 0 to 10. Higher scores indicate greater severity and more interference.
Depression | Baseline, 3 and 6 months
  Short Form 36 version 2(SF-36v2); scored from 0 (worst health) to 100 (best health)
self-efficacy | Baseline, 3 and 6 months
  general practitioner scale (GPS) to reflect specific health activities and content of Health360x Lupus. GPS response categories use a 5-point Likert scale anchored by 1 (strongly agree) and 5 (strongly disagree)
Depression | Baseline, 3 and 6 months
  Patient Health Questionnaire 9; Total scores of 5, 10, 15, and 20 represent points for mild, moderate, moderately severe and severe depression, respectively.
self-efficacy | Baseline, 3 and 6 months
  Health self-efficacy scale; A total score, on a scale of 10 to 40, or a mean scale score, on a scale of 1 to 4, can be calculated. Higher scores indicate higher perceived general self-efficacy, lower scores indicate lower perceived general self-efficacy.
Depression | Baseline, 3 and 6 months
  Patient Health Questionnaire 4; Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12). Total score ≥3 for first 2 questions suggests anxiety. Total score ≥3 for last 2 questions suggests depression.

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Pemu, MD, Principal Investigator — MSM Director of Clinical Research Center